CLINICAL TRIAL: NCT07406191
Title: Effects of Intensive Muscle Training on Cardiometabolic Risk Factors - a Randomised Controlled Study
Brief Title: WB-EMS Effects on Cardiometabolic Risk Factors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Universität Tübingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMS-KHK
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Hypertension; Metabolic Syndrome; Hypercholesterolemia; Hypertriglyceridemia; Overweight and Obesity
MeSH Terms: conditions — Hypertension; Metabolic Syndrome; Hypercholesterolemia; Hypertriglyceridemia; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Randomized controlled study with two study arms
Who Masked: Outcomes Assessor
Masking Description: The study is blinded exclusively for the measurement assistants, who do not know the status of the participant and are not permitted to ask about it.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole-body electromyostimulation (Experimental): 12 weeks of Whole-body electromyostimulation, 1.5x 20min/week
  Interventions: Other: WB-EMS
- Control group (Other): 12 weeks without additional intervention.
  Interventions: Other: Control

INTERVENTIONS:
Other: WB-EMS — 12 weeks of WB-EMS, 1.5x20 min/week
  Other Names: Electromyostimulation
  Arms: Whole-body electromyostimulation
Other: Control — 12 weeks without additional intervention and without life style changes
  Other Names: Non-intervention control group
  Arms: Control group

SUMMARY:
From the age of 50 onwards, there is a disproportionate decline in muscle strength, mass and function, which can be prevented or at least delayed by physical training. Unfortunately, many training programmes are very time-consuming and strenuous and are therefore not carried out consistently. Whole-body electromyostimulation (WB-EMS), a technology in which all major muscle groups are stimulated with an adjusted stimulation level, could be a time-effective and joint-friendly alternative.

However, there are some contraindications to the widespread use of this technology, which are particularly common in middle-aged and elderly people. For example, high blood pressure, which affects more than half of men over the age of 50 in Germany, is considered a contraindication for WB-EMS training. However, this assessment is not very reliable; at least, acute WB-EMS application does not lead to an increase in blood pressure. In addition, there are no study results available for long-term WB-EMS application in people with high blood pressure.

The present study particularly investigate whether and to what extent several weeks of WB-EMS training has an effect on resting blood pressure in people with mild blood pressure. Additionally, the effect of WB-EMS on other cardiometabolic risk factors and physical functiion will be addressed.

ELIGIBILITY:
Inclusion Criteria:

* Grade 1 hypertension: systolic 140 and/or diastolic 90 mmHg
* overweight or obese (body mass index > 25 kg/m2)

Exclusion Criteria:

* blood pressure-lowering pharmacologic therapy.
* WB-EMS application and regular resistance exercise training
* Conditions and illnesses that preclude intensive physical exertion
* Severe cardiac arrhythmia
* Heart failure
* acute pulmonary embolism
* acute myocarditis
* severe hypertension, e.g. RR > 200 mmHg systolic and/or 110 mmHg diastolic
* Contraindications for bioimpedance analysis (e.g. pacemaker)
* Contraindications for WB-EMS application (e.g. acute infections/fever, epilepsy)

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility is based on self-representation of gender identity
Enrollment: 42 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Resting blood pressure | At baseline and after 12 weeks of intervention
  Changes of mean arterial blood pressure after 10 min of rest in a sitting position as assessed by an automatic sphygmomanometer
Metabolic syndrome | At baseline and after 12 weeks of intervention
  Changes of the Metabolic Syndrome (MetS) as determined by the MetS-Z-Score according to Johnson (2007)

SECONDARY OUTCOMES:
Body fat rate | At baseline and after 12 weeks of intervention
  Changes of body fat rate as determined by Bio Impedance Analysis (BIA)
Lean body mass | At baseline and after 12 weeks of intervention
  Changes of lean body mass as determined by Bio Impedance Analysis (BIA)
Maximum muscle strength | At baseline and after 12weeks of intervention
  Changes of maximum hip-/leg extension strength as determined by a leg press
Aerobic capacity | At baseline and after 12 weeks of intervention
  Changes of aerobic capacity as determined by a stepwise crosstrainer test to submaximum exertion
Lower extremity muscle power | At baseline and after 12 weeks of intervention
  Changes of lower extremity muscle power as determined by a 5times sit to stand test
Low-level inflammation | At baseline and after 12 weeks of intervention
  Changes of inflammatory markers as determined by cytokines
Adipose-tissue derived hormones | At baseline and after 12 weeks of intervention
  Changes of adipose tissue-derived hormones as determined by adipokines
Muscle-tissue derived hormones | At baseline and after 12 weeks of intervention
  Changes of muscle-tissue derived hormones as determined by myokines
Quality of life (QoL) in people with hypertension | At baseline and after 12 weeks of intervention
  Changes in QoL in people with hypertension according to the questionnaire of Merck et al (1996]
Sleep Quality | At baseline and after 12 weeks of intervention
  Changes in sleep quality according to the Pittsburgh Sleep Quality Index questionnaire of Buysse et al. (1989)
Adverse effects | From baseline assessment to 12 week control assessment (during the intervention)
  All categories of adverse effects as determined by structured monthly telephone interview

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Kemmler, PhD, Principal Investigator — Institute of Radiology, University Hospital Erlangen, Germany
Locations (2):
- Germany (2):
  - Faculty of Medicine, University of Tuebingen, Erlangen
  - Institute of Radiology, University Hospital Erlangen, Erlangen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kemmler W, Kohl M, von Stengel S, Willert S, Kast S, Uder M. Effects of whole-body electromyostimulation with different impulse intensity on blood pressure changes in hyper- and normotensive overweight people. A pilot study. Front Physiol. 2024 Feb 22;15:1349750. doi: 10.3389/fphys.2024.1349750. eCollection 2024. PMID 38455842